CLINICAL TRIAL: NCT07103161
Title: Does a Regular Tampon or Intravaginal Pessary Mitigate Urine Leakage While Running Among Females Who Experience Exercise-induced Urinary Incontinence?
Brief Title: Managing Impact-related Leakage During Exercise Using Intravaginal Support
Acronym: MILES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Linda McLean, Full Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-06-22-8153
Record Dates: First submitted 2025-07-24; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: stress urinary incontinence; conservative treatment; pelvic floor strain; pessary; bladder support device; urinary symptoms; tampon; urine leakage; urine leakage with exercise; urine leakage with running
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Menstrual Hygiene Products

STUDY DESIGN:
Intervention Model Description: This is an assessor blind randomized crossover study design in which all participants complete a baseline visit and are then repeat the protocol at two subsequent visits, one with the tampon and one with the pessary, with the order randomized.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tampon Visit: run with tampon (Active Comparator)
  Interventions: Device: Sportex regular tampon
- Pessary Visit: run with pessary (Active Comparator)
  Interventions: Device: Uresta bladder support device

INTERVENTIONS:
Device: Uresta bladder support device — The Uresta bladder support device is an intravaginal device indicated for adult women over 18 years of age who experience stress urinary incontinence, including urine leakage during exercise and non-exercise activities such as coughing and laughing. The device is FDA-cleared and licensed by Health Canada. Participants receive the entire kit that includes the three most common sizes which fit 90% of women. Two additional sizes are available in the lab if needed. Participants will be instructed to self-insert the Uresta prior to running, following the manufacturer instructions with researcher guidance as needed. The device aims to provide mechanical support to the urethra and bladder neck to prevent urine leakage during activities that provoke leakage.
  Other Names: Uresta pessary
  Arms: Pessary Visit: run with pessary
Device: Sportex regular tampon — Participants will use a regular absorbency Sportex tampon as a conservative intravaginal support to potentially reduce stress urinary incontinence (SUI) symptoms during running. Participants will be instructed to insert the tampon prior to running into the mid-to-upper vaginal canal while standing or sitting.
  Other Names: Menstrual tampon
  Arms: Tampon Visit: run with tampon

SUMMARY:
The goal of this study is to evaluate the effectiveness of using a regular menstrual tampon or a Uresta pessary to reduce urine leakage associated with running-induced stress urinary incontinence (RI-SUI) in females aged 18 and older. Secondly, the study aims to assess whether either intervention mitigates transient changes in pelvic morphology that occur following a single running bout. Lastly, we aim to evaluate whether participants continue using either intervention during running over the 4-week period following their in-lab participation. The hypotheses are:

Hypothesis 1: Among females with RI-SUI, both a tampon and pessary used during a single running bout will reduce urinary leakage symptoms, with greater symptom reduction observed when using the pessary.

Hypothesis 2: Participants will report high satisfaction and perceived symptom improvement with both the tampon and pessary, with higher satisfaction and greater improvement reported for the pessary.

Hypothesis 3: Both the tampon and pessary will reduce pelvic floor strain incurred by the end of the run, as evidenced by less bladder neck descent, levator plate lengthening, and levator hiatus area increasing relative to that observed when no tampon or pessary is used.

Hypothesis 4: A greater proportion of participants will report continued use of the pessary compared to the tampon over the 4-week post-lab period, with higher frequency of use and fewer reported discontinuations.

We will perform within-subject comparisons against baseline values to determine the effect of each intervention on RI-SUI symptoms and pelvic organ support.

Participants will complete a baseline questionnaire to collect demographic information and assess incontinence severity. They will then attend three laboratory visits within a 10-day period. At each visit, bladder volume will be standardized to between 100 and 200mL, then the participant will undergo three-dimensional (3D) transperineal ultrasound imaging conducted in a standing position. Following imaging, participants will complete a treadmill protocol consisting of 25-minutes running at a moderately difficult pace (rated at 13 - 14 on the Borg Perceiver Rate of Exertion scale), followed by 5 minutes of running at a higher intensity pace. During the run, participants will be asked at 5 minute intervals whether they experienced any urine leakage and to report their perceived amount of leakage. The ultrasound image protocol will be repeated immediately after the run.

Participants will be allowed to keep the pessary and will be contacted 4-weeks after the final visit to evaluate whether or not they continued use of a tampon or the pessary, and, if so, we will ask them to report their satisfaction with the intervention(s) they used.

DETAILED DESCRIPTION:
More than 30% of females experience urinary incontinence (UI) during exercise. For many women, urine leakage during exercise can become a barrier to staying active, leading them to modify their exercise routine or avoid triggering activities altogether. Beyond the physical inconvenience, urinary incontinence can affect self-esteem, social participation, and mental health. Helping women stay active without embarrassment or fear of leakage has both physical and psychological benefits.

The pelvic floor muscles (PFMs) and associated connective tissues play a critical role in continence control. These structures support the pelvic organs and help maintain their positioning such that the urethra is optimally compressed during increases in intra-abdominal pressure. Dysfunction of the PFMs and connective tissues will cause the bladder to descend during weight-bearing activities, and the urethra, no longer in its optimal position, may remain open - resulting in urine leakage. This form of UI, known as stress urinary incontinence (SUI), is commonly experienced as urine leakage during tasks such as coughing, laughing, and physical activity. High-impact movements like running, jumping, and inclined walking are known to increase the loads experienced by the pelvic floor, making SUI especially common during these types of activities.

Intravaginal products such as tampons and pessaries (reusable medical devices placed in the vagina) are recommended to help manage UI during everyday activities such as coughing and sneezing. However, their effectiveness during physical activities - such as running or brisk walking - remains unclear. This study aims to determine whether a standard menstrual tampon and/or a bladder support (Uresta) pessary can reduce urine leakage during running and/or brisk walking in active females. A secondary objective is to assess whether these devices mitigate the descent of the bladder that we have observed in females after running or brisk walking. Lastly, we aim to assess continued device use over a 4-week period following all laboratory visits.

By evaluating the effectiveness of accessible, non-invasive devices, this research may offer immediate, low-barrier strategies to help active women self-manage urinary incontinence - empowering them to maintain their physical activity routines and support their long-term health.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age
* Participate in any exercise or sport modality involving running or brisk walking
* Experiences urine leakage during running or brisk walking
* Speak and read English or French

Exclusion Criteria:

* No urine leakage in the first laboratory assessment (baseline / no intervention)
* Currently pregnant or have been pregnant in the previous 6 months
* Had or have had cardiac, pulmonary, metabolic and/or neurological conditions
* History of incontinence surgery
* Hysterectomy
* Symptoms consistent with urgency incontinence only
* Experience pain with tampon use or during gynecologic examinations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Urine leakage severity | At Baseline (Visit 1), and at Visit 2 and Visit 3, which will occur within 10 days of Baseline.
  Self-reported urine leakage is evaluated as presence (yes/no) and amount (drops, squirts, gush) every 5 minutes during a 38-minute treadmill run. Leakage severity index is calculated as the proportion of 5-minute blocks with leakage times the median leakage amount per block.

SECONDARY OUTCOMES:
Participant's perception of improvement | At Visit 2 and Visit 3 only, which will occur within 10 days of Baseline (Visit 1).
  Participants report perception of improvement with each device on a scale of 0% (not improved) to 100% (very much improved).
Change in levator plate length observed after an acute running bout | At Baseline (Visit 1), Visit 2, and Visit 3 - each with pre- and post-running assessments, within 10 days of Baseline.
  Levator plate length will be assessed before and after running under each condition. The primary outcome is the change in levator plate length, calculated as the difference between pre- and post-run measurements. Levator plate length is measured using 2D transperineal ultrasound imaging of the pelvic structures, acquired with participants in the standing position. The measurement is defined as the straight-line distance between the anorectal junction and the pubic symphysis.
Change in bladder neck height observed after an acute running bout | At Baseline (Visit 1), Visit 2, and Visit 3 - each with pre- and post-running assessments, within 10 days of Baseline.
  Bladder neck height will be assessed before and after running under each condition. The primary outcome is the change in bladder neck height, calculated as the difference between per- and post-run measurements. Bladder neck height is measured using 2D transperineal ultrasound imaging of the pelvic structures, acquired with participants in the standing position. The measurement is defined as the perpendicular distance from the pubic symphyseal line to the bladder neck.
Change in levator hiatus area observed after an acute running bout | At Baseline (Visit 1), Visit 2, and Visit 3 - each with pre- and post-running assessments, within 10 days of Baseline.
  Levator hiatus area will be assessed before and after running under each condition. The primary outcome is the change in levator hiatus area, calculated as the difference between pre- and post-run measurements. Levator hiatus area is measured using 3D transperineal ultrasound imaging of the pelvic structures, acquired with participants in the standing position. The measurement is defined as the hypoechoic region visualized in the transverse plane.
Use of tampon or pessary throughout the 4-week post-lab period | At 4-week follow-up (4 weeks after Visit 3, approximately Day 38 post-Baseline).
  Participants complete an online questionnaire that evaluates their use of either the tampon or pessary intervention during running over a 4-week period after completing the in-lab component of the study. They are asked whether they used the tampon or pessary while running (Yes/No) and to rate the frequency of usage on a scale of 0 (not used) to 100 (used during every run). If they did not use the pessary/tampon at all or if they stopped using the pessary/tampon during the 4-week period, they are asked to share the number of runs they ran with the device and their reasons for stopping its usage.

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, PhD., Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Faculty of Health Sciences building, 200 Lees Avenue, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared to investigators who contact the researchers and request access.
Supporting Information: Study Protocol, SAP
Time Frame: Information will be available beginning 1 month after publication with no end date.
Access Criteria: No data sharing agreement necessary. Data will be made available to researchers wishing to perform secondary analyses or include the data in systematic reviews or meta-analyses.

REFERENCES:
- [Background] Raizada V, Mittal RK. Pelvic floor anatomy and applied physiology. Gastroenterol Clin North Am. 2008 Sep;37(3):493-509, vii. doi: 10.1016/j.gtc.2008.06.003. PMID 18793993
- [Background] Petter Rodrigues M, Berube ME, Charette M, McLean L. Conservative interventions for female exercise-induced urinary incontinence: a systematic review. BJU Int. 2024 Dec;134(6):906-917. doi: 10.1111/bju.16474. Epub 2024 Jul 23. PMID 39043585
- [Background] Lovatsis D, Best C, Diamond P. Short-term Uresta efficacy (SURE) study: a randomized controlled trial of the Uresta continence device. Int Urogynecol J. 2017 Jan;28(1):147-150. doi: 10.1007/s00192-016-3090-9. Epub 2016 Jul 20. PMID 27438055
- [Background] Leitner M, Moser H, Eichelberger P, Kuhn A, Baeyens JP, Radlinger L. Evaluation of pelvic floor kinematics in continent and incontinent women during running: An exploratory study. Neurourol Urodyn. 2018 Feb;37(2):609-618. doi: 10.1002/nau.23340. Epub 2017 Jul 4. PMID 28675537
- [Background] Farrell SA, Baydock S, Amir B, Fanning C. Effectiveness of a new self-positioning pessary for the management of urinary incontinence in women. Am J Obstet Gynecol. 2007 May;196(5):474.e1-8. doi: 10.1016/j.ajog.2006.11.038. PMID 17466709
- [Background] Falah-Hassani K, Reeves J, Shiri R, Hickling D, McLean L. The pathophysiology of stress urinary incontinence: a systematic review and meta-analysis. Int Urogynecol J. 2021 Mar;32(3):501-552. doi: 10.1007/s00192-020-04622-9. Epub 2021 Jan 8. PMID 33416968
- [Background] Dakic JG, Hay-Smith J, Cook J, Lin KY, Calo M, Frawley H. Effect of Pelvic Floor Symptoms on Women's Participation in Exercise: A Mixed-Methods Systematic Review With Meta-analysis. J Orthop Sports Phys Ther. 2021 Jul;51(7):345-361. doi: 10.2519/jospt.2021.10200. Epub 2021 May 10. PMID 33971737
- [Background] Berube ME, McLean L. The acute effects of running on pelvic floor morphology and function in runners with and without running-induced stress urinary incontinence. Int Urogynecol J. 2024 Jan;35(1):127-138. doi: 10.1007/s00192-023-05674-3. Epub 2023 Nov 22. PMID 37991566
- [Background] Waetjen LE, Subak LL, Shen H, Lin F, Wang TH, Vittinghoff E, Brown JS. Stress urinary incontinence surgery in the United States. Obstet Gynecol. 2003 Apr;101(4):671-6. doi: 10.1016/s0029-7844(02)03124-1. PMID 12681869
- [Background] Serdar CC, Cihan M, Yucel D, Serdar MA. Sample size, power and effect size revisited: simplified and practical approaches in pre-clinical, clinical and laboratory studies. Biochem Med (Zagreb). 2021 Feb 15;31(1):010502. doi: 10.11613/BM.2021.010502. Epub 2020 Dec 15. PMID 33380887
- [Background] Shaw JM, Hamad NM, Coleman TJ, Egger MJ, Hsu Y, Hitchcock R, Nygaard IE. Intra-abdominal pressures during activity in women using an intra-vaginal pressure transducer. J Sports Sci. 2014;32(12):1176-85. doi: 10.1080/02640414.2014.889845. Epub 2014 Feb 28. PMID 24575741
- [Background] Rzymski P, Burzynski B, Knapik M, Kociszewski J, Wilczak M. How to balance the treatment of stress urinary incontinence among female athletes? Arch Med Sci. 2020 Oct 21;17(2):314-322. doi: 10.5114/aoms.2020.100139. eCollection 2021. PMID 33747266
- [Background] Nygaard I, Girts T, Fultz NH, Kinchen K, Pohl G, Sternfeld B. Is urinary incontinence a barrier to exercise in women? Obstet Gynecol. 2005 Aug;106(2):307-14. doi: 10.1097/01.AOG.0000168455.39156.0f. PMID 16055580
- [Background] Nekkanti S, Wu JM, Hundley AF, Hudson C, Pandya LK, Dieter AA. A randomized trial comparing continence pessary to continence device (Poise Impressa(R)) for stress incontinence. Int Urogynecol J. 2022 Apr;33(4):861-868. doi: 10.1007/s00192-021-04967-9. Epub 2021 Sep 9. PMID 34505171
- [Background] Imamura M, Williams K, Wells M, McGrother C. Lifestyle interventions for the treatment of urinary incontinence in adults. Cochrane Database Syst Rev. 2015 Dec 2;2015(12):CD003505. doi: 10.1002/14651858.CD003505.pub5. PMID 26630349
- [Background] Goldstick O, Constantini N. Urinary incontinence in physically active women and female athletes. Br J Sports Med. 2014 Feb;48(4):296-8. doi: 10.1136/bjsports-2012-091880. Epub 2013 May 18. PMID 23687004
- [Background] Duenas-Garcia OF, Shapiro RE, Gaccione P. Safety and Efficacy of a Disposable Vaginal Device for Stress Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2021 Jun 1;27(6):360-364. doi: 10.1097/SPV.0000000000000861. PMID 32453209
- [Background] Chisholm L, Delpe S, Priest T, Reynolds WS. Physical Activity and Stress Incontinence in Women. Curr Bladder Dysfunct Rep. 2019 Sep;14(3):174-179. doi: 10.1007/s11884-019-00519-6. Epub 2019 Jul 1. PMID 31456864
- [Background] Brown WJ, Miller YD. Too wet to exercise? Leaking urine as a barrier to physical activity in women. J Sci Med Sport. 2001 Dec;4(4):373-8. doi: 10.1016/s1440-2440(01)80046-3. PMID 11905931
- [Background] Brennand E, Ruiz-Mirazo E, Tang S, Kim-Fine S; Calgary Women's Pelvic Health Research Group. Urinary leakage during exercise: problematic activities, adaptive behaviors, and interest in treatment for physically active Canadian women. Int Urogynecol J. 2018 Apr;29(4):497-503. doi: 10.1007/s00192-017-3409-1. Epub 2017 Jul 6. PMID 28685262
- [Background] Bo K. Urinary incontinence, pelvic floor dysfunction, exercise and sport. Sports Med. 2004;34(7):451-64. doi: 10.2165/00007256-200434070-00004. PMID 15233598
- [Background] Al-Shaikh G, Syed S, Osman S, Bogis A, Al-Badr A. Pessary use in stress urinary incontinence: a review of advantages, complications, patient satisfaction, and quality of life. Int J Womens Health. 2018 Apr 17;10:195-201. doi: 10.2147/IJWH.S152616. eCollection 2018. PMID 29713205